CLINICAL TRIAL: NCT06304363
Title: Braining Study - Physical Exercise in Psychiatry - Evaluation of Acute Effects
Brief Title: Braining - Evaluation of Acute Effects of Physical Exercise
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Braining booster
Record Dates: First submitted 2024-02-23; First posted 2024-03-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Psychiatric Disorder
Keywords: Psychiatric disorder; Physical Exercise
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity (Experimental): Patients are encouraged to participate in physical exercise at the psychiatric unit
  Interventions: Behavioral: Braining

INTERVENTIONS:
Behavioral: Braining — "Braining" is a clinical invention that helps patients in psychiatry to start and execute physical exercise (PE) regularly in psychiatric care. The core components are basic moderate to vigorous aerobic group training session and motivational work led by the psychiatric staff. Braining is used as add-on treatment to regular psychiatric care and is included in the patient care plan.

SUMMARY:
"Braining" is a clinical method for physical exercise as adjunctive therapy in psychiatric care. The core components are personnel-led group training sessions and motivating contact with psychiatric staff, as well as measurements and evaluations before and after a training period.

The scientific purpose of this study is to investigate immediate and short-term effects of a booster-session of several Braining classes.

DETAILED DESCRIPTION:
"Braining" is a clinical invention that helps patients in psychiatry to start and execute physical exercise (PE) regularly in psychiatric care. The core components are basic moderate to vigorous aerobic group training sessions and motivational work led by the psychiatric staff. Braining is used as add-on treatment to regular psychiatric care and is included in the patient care plan.

In the present study, the focus is on the acute effects of a booster session of one to three Braining classes on psychiatric symptoms and biomolecular markers as well as impact on motivational factors.

Participants are recruited from the final cohort (N = 51) of the previous retrospective study, (Physical Exercise as Adjunctive Therapy for Affective Disorder and Anxiety).This final cohort will be contacted to give written consent to partake in the booster session. The Braining classes each have a duration of 30 minutes and are scheduled over the course of a week.

Descriptive data on participating patients will be collected before the booster week. This will include age, gender, diagnoses, employment status. In conjunction with this, basic psychiatric and somatic examinations will be conducted.

During each Braining class, participants' activity level will be measured with a heart rate monitor to ascertain achieving moderate to vigorous intensity. Directly before and after each class, current anxiety level will be measured on a Visual Analogue Scale 0-100.

Within 30 minutes before and after one Braining class, venous blood samples (50 ml) will be taken for biomolecular markers. Blood samples include 1) inflammation markers such as high-sensitivity C-reactive protein hsCRP, 2) Brain-derived neurotrophic factor BDNF, 3) telomerase activity and 4) epigenetic markers.

Before and after the booster week, self-assessments scales for anxiety and depressive symptoms will be administered. Qualitative data on participants' experience as well as motivational factors will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Included in the retrospective study Physical Exercise as Adjunctive Therapy for Affective Disorder and Anxiety and has given informed consent to participation in a Braining booster session.

Exclusion Criteria:

* Severe psychiatric disorder such as mania and psychosis
* Medical conditions such as heart- and lung diseases where PE is contraindicated.
* Unable to understand written and spoken Swedish language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety Visual Analogue Scale (VAS) | Pre- to post-exercise class, timeframe 2 hours
  Self-rated anxiety levels on a scale from 0 to 100, where 0 is no anxiety and 100 is maximal anxiety.

SECONDARY OUTCOMES:
Beck Anxiety Inventory BAI | Pre-intervention to post-intervention, timeframe 1 week
  Self-report measure of anxiety during the last week. 21 items, score ranges from 0 to 63 with higher scores indicating more severe anxiety symptoms.
Montgomery-Åsberg Depression Rating Scale MADRS | Pre-intervention to post-intervention, timeframe 1 week
  Clinician-rated scale to assess degree of depressive symptoms. 10 items. Minimum value 0 and maximum value 60, where higher values indicate more depressive symptoms.
High sensitivity C-reactive protein hsCRP | Pre- to post-exercise class, timeframe 2 hours
  Blood marker of inflammation and infection, mmol/L
Brain-derived neurotrophic factor BDNF | Pre- to post-exercise class, timeframe 2 hours
  Stimulates and controls neurogenesis
Telomerase activity | Pre- to post-exercise class, timeframe 2 hours
  Enzyme activity in blood
Motivational factors of continued exercise | Pre-intervention to post-intervention, timeframe 1 week
  Semi-structured interview derived from motivational interviewing

CONTACTS AND LOCATIONS:
Overall Officials: Lina Martinsson, Principal Investigator — Karolinska Institutet
Locations (1):
- Region Stockholm, Psykiatri Sydväst (Psychiatric Clinic Psychiatry Southwest), Stockholm, Stockholm County, Sweden